CLINICAL TRIAL: NCT06275464
Title: A Phase 1, 2-Part, Randomized, Double-Blind, Placebo Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BT-600 Single and Multiple Ascending Oral Doses in Healthy Adult Subjects
Brief Title: BT-600 Single and Multiple Ascending Oral Doses in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biora Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BT-600-101
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (8):
- 5mg SAD (Active Comparator)
  Interventions: Combination Product: BT-600
- 5mg SAD placebo (Placebo Comparator)
  Interventions: Combination Product: BT-600 Placebo
- 10mg SAD (Active Comparator)
  Interventions: Combination Product: BT-600
- 10mg SAD placebo (Placebo Comparator)
  Interventions: Combination Product: BT-600 Placebo
- 5mg MAD (Active Comparator)
  Interventions: Combination Product: BT-600
- 5mg MAD placebo (Placebo Comparator)
  Interventions: Combination Product: BT-600 Placebo
- 10mg MAD (Active Comparator)
  Interventions: Combination Product: BT-600
- 10mg MAD placebo (Placebo Comparator)
  Interventions: Combination Product: BT-600 Placebo

INTERVENTIONS:
Combination Product: BT-600 — NaviCap device containing liquid formulation of Tofacitinib
  Arms: 10mg MAD; 10mg SAD; 5mg MAD; 5mg SAD
Combination Product: BT-600 Placebo — NaviCap device containing placebo formulation
  Arms: 10mg MAD placebo; 10mg SAD placebo; 5mg MAD placebo; 5mg SAD placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 1 study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of BT-600 when administered in single and multiple ascending doses to healthy participants. The study will enroll up to 48 participants, with participation lasting 2-3 weeks in addition to up to 28 days (about 4 weeks) for screening.

The purposes of this study are to learn about the safety and tolerability of single and multiple rising oral doses of BT-600, assess the blood and tissue levels of tofacitinib released from BT-600, and assess the body's effects to the study drug following oral doses of BT-600 in blood and tissue in healthy adult participants.

BT-600 is a swallowable drug/device combination product designed to deliver a liquid formulation of tofacitinib to the colon and dispense the study drug throughout the colon. BT-600 consists of two components, the drug part containing a reservoir, which will be filled with liquid tofacitinib, and the drive part. The drive part contains the hardware and software that identifies the colon region and then dispenses the drug to the specific region. The device which contains the drug is referred to as the NaviCap™ device. The NaviCap device is approximately the size of a fish oil pill, is made of plastic material known to be safe for ingestion and has rounded ends for ease of swallowing. Liquid tofacitinib in the reservoir is automatically released when the BT-600 localization technology determines that it has reached the colon. BT-600 passes through the colon and the NaviCap device is excreted via a bowel movement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult male or female, 19-50 years of age.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, or vital signs, as deemed by the Investigator or designee.
* Laboratory results within normal range or not clinically significant as determined by the Investigator at Screening.
* Understands the study procedures in the informed consent form (ICF) and willing and able to comply with the protocol.

Exclusion Criteria:

* History of any illness, clinically significant medical condition, or disease, that in the opinion of the Investigator or designee might confound the results of the study or pose an additional risk to the subject by participation in the study.
* Major surgery within 4 weeks before study entry or anticipated during the study period.
* Has clinically significant active infectious disease or history of significant infectious disease.
* Participation in another clinical study within 30 days prior to the first dosing or five half-lives of the Investigational Product tested, whichever is longer. The window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.
* Female subjects with a positive pregnancy test at the Screening visit or at Check-in, or who are lactating.
* Donation of blood or significant blood loss within 56 days prior to the first dosing.
* Plasma donation within 7 days prior to the first dosing.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 2 weeks
  Number of Treatment-Emergent Adverse Events.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Assessments | Up to 7 days
  Maximum Plasma Concentration [Cmax] at Days 1, 2, 3, 4, 5, 6, 7.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Leader, Study Director — Biora Therapeutics, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No